CLINICAL TRIAL: NCT04444076
Title: Clinical Trial on the Effect of REGENETEN Bioinductive Implant in the Supraspinatus Tendon Repair
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MALLAMANGUITO
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Supraspinatus Tear
Keywords: Supraspinatus Tear; REGENETEN

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REGENETEN Bioinductive Implant (Experimental): REGENETEN bioinductive Implant,a bovine mesh that will be implanted following supraspinatus tendon repair.
  Interventions: Device: REGENETEN Bioinductive Implant
- Standard of Care (No Intervention): Supraspinatus tendon repair.

INTERVENTIONS:
Device: REGENETEN Bioinductive Implant — REGENETEN bioinductive Implant,a reconstituted bovine origin type I collagen mesh with a proprietary high porosity system that is commercialized sterile, dehydrated and desiccated in two sizes (20x26mm and 25x31mm). It will be implanted following supraspinatus tendon repair.
  Arms: REGENETEN Bioinductive Implant

SUMMARY:
This study aims a determine the effect that the addition of REGENETEN Bioinductive Implant has on Supraspinatus Tendon Repair. 120 patients will be included in this prospective, randomized, parallel group study.

DETAILED DESCRIPTION:
The rotator cuff tear is one of the most frequent pathologies in the shoulder joint. When there are many symptoms these breaks are repaired surgically. The success rate of healing of these injuries is between 30% and 80%. In two recent studies conducted at two of the centers participating in this trial, the success rate of repair was 75% (unpublished data) and 70% respectively.

The use of high porosity resorbable bovine collagen meshes as bioinductive scaffolds for cuff repair seems to be a valid alternative when trying to improve the success rate in the healing of rotator cuff injuries.

REGENETEN Bioinductive Implant (a high porosity reconstituted type I collagen mesh of bovine origin) is applied to the repaired tendon. In a pilot study of 9 subjects with full thickness supraspinatus ruptures who underwent tendon repair and subsequently had the implant associated with the rupture, a significant clinical improvement was observed after one year and was observed on magnetic resonance imaging ( RM) 100% healing of breaks. In a study of 33 subjects with partial thickness tears treated with the implant alone, improvement in MRI characteristics of the tendon was observed in 31 cases. There is a study that performs a histological analysis of samples obtained in 7 subjects in whom the implant was used. No evidence of foreign body reaction or inflammatory reaction was observed. In none of the three studies where said implant was used in humans were any complications or adverse effects related to the use of said implant observed.

The objective of the study is to evaluate the effect that the addition of REGENETEN bovine collagen mesh has on tendon repair on MRI performed one year after surgery.

The study does not in itself pose a greater risk than the usual practice for the patient, since in these subjects where the implant could be used as a supplement to the repair, having already obtained the CE marking.

ELIGIBILITY:
Inclusion Criteria:

* Patients who, after having received information about the design, the purposes of the study, the possible risks that may arise from it, and who may at any time deny their collaboration, give their written consent to participate in the study.
* >18 years
* Patients who present:

  * Symptomatic ruptures of the supraspinatus muscle (SE) with or without involvement of the infraspinatus (IE) with anteroposterior size of the rupture of 1 to 4 cm.
  * With less than 3cm of retraction,
  * With the absence of severe muscular atrophy confirmed by magnetic resonance imaging or CT (Absence of Goutalier grade I or II atrophy in muscle mass). MRI or CT must have been performed at most 6 months before the intervention.
  * That it be confirmed during the exploratory arthroscopy at the beginning of the intervention.
  * That after repair a coverage of the native footprint of the tendon of at least 80% is obtained
* No presence of rupture that requires repair in the tendons of the subscapularis muscles or minor round
* Understand the purpose of the study and be available for regular hospital visits.
* Negative urine pregnancy test performed in the 7 days prior to the start of study treatment in premenopausal women or <2 years after menopause

Exclusion Criteria:

* Pregnancy or planning to become pregnant during the course of the study.
* SE tendon tears of more than 3cm retraction
* Tendon ruptures of the SE and IE muscles with anteroposterior size of the rupture greater than 4 cm.
* SE and / or IE tendon ruptures that are considered irreparable or only partially repairable at the time of the intervention
* Presence of ruptures of the subscapularis and / or minor round tendons
* Presence of grade III or IV Goutallier atrophy in the supraspinatus muscle mass
* History of other orthopedic pathologies in the affected shoulder (previous shoulder surgeries, fractures, tendon re-ruptures of the supraspinatus or other tendons, rheumatic diseases, septic arthritis, ...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Integrity of the tendon repaired in an MRI study one year after the intervention using the Sugaya classification (Sugaya H (2005)). | 12 months
  This is a classification system described by Sugaya et al. which uses magnetic resonance imaging in order to evaluate tendon integrity after rotator cuff repair. Postoperative cuff integrity is classified into 5 categories: type I, sufficient thickness with homogenously low intensity; type II, sufficient thickness with partial high intensity; type III, insufficient thickness without discontinuity; type IV, presence of minor discontinuity; type V, presence of major discontinuity

SECONDARY OUTCOMES:
Change in pain levels. Measured with questions 3 to 6 of the Brief Pain Inventory. | 3 months, 6 months and 12 months after surgery
  This item has a scale of 0 to 10 with 0 indicating "No pain" and 10 indicating "Pain as bad as you can imagine"
Functional changes, measured with the Constant-Murley Scale. | 3 months, 6 months and 12 months after surgery.
  The Constant-Murley Shoulder Score is a scoring method used by clinicians to assess function of the shoulder. The score is on a scale of 0 to 100, with 0 being no shoulder function and 100 being excellent function.
Functional changes, measured with ASES questionnaire. | 3 months, 6 months and 12 months after surgery.
  The American Shoulder and Elbow Surgeons (ASES) questionnaire was developed to provide a standardized method for evaluating shoulder function and has been validated in patients with any array of shoulder pathologies. The range is from 0 to 100, with 0 being worst, and 100 being best.
Changes in quality of life measured with EQ-5D-5L questionnaire. | 3 months, 6 months and 12 months after surgery.
  The Euro Quality of Life Five Dimensions 5 Level (EQ-5D-5L) questionnaire consists of two parts: a descriptive system and a Visual Analogue Scale.
  The descriptive system describes the health state and consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Patients who reported problems were then categorized into two categories, a "has no problem" category (health state code of 1) and "has problem" category (health state code of 2-5) for each level of each dimension.
  The second part of the EQ-5D-5L questionnaire is the EQ-VAS, which is a thermometer-like scale (ranging from 0 to 100) that reflects the patient's health in general. EQ-VAS represents the patient perspective, where 0 indicates the worst imaginable health state and 100 reflects the best imaginable health state.
Number of patients with complications in both arms | 12 months
  Rate of complications, including: infection, implant intolerance, readmission, reoperation, or fracture.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Ruiz Iban, MD, PhD, Principal Investigator — Hospital Ramón y Cajal, Spain
Locations (1):
- Hospital Ramón y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No